CLINICAL TRIAL: NCT06886178
Title: The Effect of the STIL Orthosis on Action Tremor Severity in People With Parkinson's Disease
Brief Title: Effectiveness of STIL Orthosis in PD
Acronym: STIL-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: The Dutch Brain Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL86972.091.24
Record Dates: First submitted 2025-03-03; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Parkinson&Amp;#39;s Disease; Action Tremor
Keywords: Parkinson's disease; Action tremor; Orthosis
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baseline-Intervention-Sham (Experimental): Order of tremor assessments: Baseline > STIL Orthosis > Sham
  Interventions: Device: STIL Orthosis; Device: Sham
- Baseline-Sham-Intervention (Experimental): Order of tremor assessments: Baseline > Sham > STIL Orthosis
  Interventions: Device: STIL Orthosis; Device: Sham

INTERVENTIONS:
Device: STIL Orthosis — STIL Orthosis, a brace for the arm equipped with passive dampening designed to suppress high-frequency movements.
Device: Sham — A version of the STIL Orthosis that is visually indistinguishable from original, but which does not have the passive dampening mechanism.

SUMMARY:
Parkinson's disease is a neurodegenerative condition that leads to uncontrollable shaking (tremor), which can substantially impair everyday activities. The goal of this clinical trial is to learn if the STIL Orthosis works as a treatment option for tremor in people with Parkinson's disease. The main questions it aims to answer are:

* Does the STIL Orthosis reduce tremor?
* Are users satisfied with the usability and comfort of the STIL Orthosis?
* Does the STIL Orthosis have any adverse effects?

Participants' tremor will be measured during three conditions:

* While wearing the STIL Orthosis
* While wearing an orthosis without dampening (sham)
* While wearing no orthosis (baseline)

Researchers will compare the severity of tremor while wearing the STIL Orthosis against tremor during sham and baseline.

DETAILED DESCRIPTION:
* <b>Background</b>: Tremor is a common symptom in people with Parkinson's disease (PD), affecting 75% of patients. While PD tremor usually occurs at rest, 46-93% of patients also have action tremor. Action tremor often does not respond to dopaminergic medication, and stereotactic surgery is invasive and unsuitable for many patients. By interfering with daily activities, action tremor can reduce independence and quality of life, necessitating new treatments.
* <b>STIL Orthosis</b>: The STIL Orthosis, a CE-certified device, aims to reduce tremor by dampening wrist flexion-extension and forearm pronation-supination. It features dampeners that limit high-frequency movements, such as tremor, while maintaining voluntary movements. In patients with essential tremor (n=24), the STIL Orthosis reduced action tremor severity during daily activities by 65-87% compared to baseline. This suggests that it could be a promising treatment for PD action tremors.
* <b>Design</b>: In this study, 25 PD patients will be recruited to test whether the STIL Orthosis can be used to treat PD-related action tremor. Action tremor will be measured under three conditions: while wearing the STIL Orthosis (intervention), while wearing an orthosis without dampening (sham), and while wearing no orthosis (baseline). Severity of action tremor in all conditions will be assessed using the TETRAS scale.
* <b>Primary outcome</b>: The primary outcome of this study is action tremor severity, measured using the <b>TETRAS scale</b>. The main study endpoint is the <b>difference in TETRAS scores between two conditions (intervention vs. sham and intervention vs. baseline)</b>.
* <b>Secondary outcomes</b>: As secondary outcomes, we will measure tremor severity using the MDS-UPDRS part III scale, focusing on items related to postural, kinetic, and rest tremor (3.15, 3.16, 3.17). We will also measure tremor power using surface electromyography (sEMG) and accelerometry. Furthermore, we will assess perceived change in tremor using the PGC-I, user satisfaction on relevant items from the D-QUEST, and product safety using an adverse events report form.
* <b>Sample size calculation</b>: The sample size calculation is based on a pilot study with 8 Parkinson's disease patients experiencing action tremor in the forearm, which showed an effect size of 1.24 1.86 for MDS-UPDRS part 3 (tremor items 3.15, 3.16, and 3.17) and 2.21 for TETRAS. Given that patients only benefit from a device that has a large effect on their tremor, an effect size <b>Cohen's d=0.8</b> was chosen, which is also common practice in the medical literature. In total, two main comparisons will be done on the primary outcome (TETRAS score): intervention vs. sham, intervention vs. baseline. To adjust for multiple statistical tests, a Bonferroni correction of <b>alpha = 0.05/2 = 0.025</b> is used. To achieve <b>80% power in a two-sided paired t-test</b>, a minimum of <b>18 patients</b> needs to be included. In order to compensate for possible drop-outs, 25 patients will be included for this clinical investigation.
* <b>Statistical analysis</b>: All analyses will follow the intention-to-treat principle. Paired-samples t-test will be used to test for intervention-related effects on action tremor severity. In the event that tremor severity scores are not normally distributed, Wilcoxon signed rank tests will be used instead.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years of age.
* Willing to sign the informed consent.
* Diagnosed with Parkinson's disease by a neurologist or movement disorders specialist.
* Action tremor in one or two arms (clinical severity score of at least 2 on their dominant side, on MDS-UPDRS items 3.15 or 3.16).
* At least experiencing wrist flexion/extension or forearm pronation/supination tremor.

Exclusion Criteria:

* Diagnosed with any other neurological disorder, such as epilepsy, Essential tremor, functional tremor, physiologic tremor, cerebellar tremor, MS, spasticity, ataxia, dystonia, Alzheimer's disease or dementia, atypical parkinsonism, peripheral neuropathy affecting the arms (e.g., carpal tunnel syndrome).
* Disease duration of >= 7 years.
* Using a high dose of dopamine agonists, i.e., a levodopa equivalent dose (LED) of >150 mg for agonists, equivalent to approximately 1.5 mg pramipexole and 5 mg rotigotine). This is done, because dopamine agonists can have longer-lasting effects beyond 12 hours after the last dose (which is our criterion for OFF, to ensure feasibility for participants). If patients take higher doses of dopamine agonists, they may still be *ON* at the time of study.
* Experiencing severe bradykinesia/rigidity, to such an extent that the participant is unable to perform the ADL tasks (drinking, eating, pouring water).
* Limited movement or muscle function in the arm/hand (for contractures or muscle diseases), or loss of muscle function in one arm (e.g., due to paralysis, or amputation).
* Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin on the forearm or hand that would wear the orthosis during the clinical investigation.
* Consuming excessive alcohol (more than 21 glasses per week for men and 14 glasses per week for women), as defined in the GGZ guidelines on alcohol use.
* Having received a botulinum toxin injection to suppress hand tremor in the past six months, or planned in the coming 60 days.
* Previous or planned Deep Brain Stimulation (DBS) at time of study enrollment that interferes with testing.
* Change in any tremor medication in the past 30 days or planned during the period of testing.
* A hand circumference smaller than 170 mm, or larger than 250 mm.
* An upper arm circumference smaller than 180 mm, or larger than 350 mm.
* Patch/band-aid allergies.
* Participant is unable to communicate with the investigator and staff due to: (1) not mastering the Dutch and English language, (2) blindness, (3) deafness, (4) illiteracy.
* Pregnancy or anticipated pregnancy at time of study enrollment.
* Any health condition that in the neurologist's opinion should preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
TETRAS | Day 1
  Tremor severity is assessed using the Tremor Research Group Essential Tremor Rating Scale (TETRAS), which is a validated scale specifically designed for essential tremor, the most common action tremor worldwide.
  TETRAS will be rated by two independent assessors, based on a video recording. The scale covers 7 postural and kinetic tasks (postural outstretched arms, postural wing beating, finger-to-nose maneuver, eating, drinking, pouring, Archimedes spiral), which are selected to accurately represent the difficulties that PD patients experience with per-forming ADL tasks. A TETRAS score is rated on the baseline, and for the sham and STIL Orthosis conditions. Tremor is rated on a 0 to 4 scale per task, with 0 indicating no visible tremor and 4 indicating a tremor with an amplitude exceeding 20 cm. Combining the 7 tasks from the TETRAS scale, a maximum sum score of 28 points can be achieved per condition.

SECONDARY OUTCOMES:
MDS-UPDRS part III tremor items | Day 1
  Tremor severity is also assessed using the MDS-UPDRS part III scale. Items 15, 16, and 17, of the MDS-UPDRS part III for postural, kinetic, and rest tremor will be used for assessment of the arm, respectively. Tremor is rated on a 5-point scale, with 0 indicating no tremor and 4 indicating a tremor with an amplitude of at least 10 cm. Note that the tasks for this rating are distinct from the TETRAS scale.
Tremor power | Day 1
  Quantification of tremor power will be based on movement data from accelerometry and using surface electromyography (sEMG). Again, the same 7 tasks (postural out-stretched arms, postural wing beating, finger-to-nose manoeuvre, eating, drinking, pour-ing, Archimedes spiral) and resting posture are used to compare baseline, sham and in-tervention conditions. Tremor power is obtained through signal processing.
PGI-I | Day 1
  Perceived change in tremor while wearing the sham and STIL Orthosis, using the Patient Global Impression of Improvement (PGI-I) scale. This questionnaire is a single-item scale that measures a patient's perception of improvement or deterioration in their condition following treatment. Answers range from 'very much improved' to 'very much wors-ened'.
D-QUEST | Day 1
  User satisfaction is evaluated with a subset of the Dutch Quebec User Evaluation of Satisfaction with Assistive Technology (D-QUEST) (Demers et al., 2001 & 2002). This questionnaire consists of 8 questions regarding comfort and usability of the device itself and 5 questions about the service of the manufacturer. Only 4 questions about satisfaction of the device itself will be questioned. Satisfaction is measured on a 1-5 scale, ranging from 'completely not satisfied' to 'very satisfied'. Additional questions regarding comfort will be asked to examine possible adverse-effects more detailed.
Adverse events | Day 1
  Product safety will be assessed using the Dutch version of NCCIH's Adverse Events Report Form. This form is used to report the severity, relationship to the study, taken action, outcome of the (S)AE and whether it was expected or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Donders Institute for Brain, Cognition and Behaviour, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other research sites upon approval of reasonable requests.